CLINICAL TRIAL: NCT02994225
Title: Axillary Reverse Mapping Using Near-infrared Imaging in Invasive Breast Cancer: Predictors of Nodal Positivity
Acronym: ARMONIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A01623-48; 2016/2462 (Other: CSET number)
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Subcutaneous injection (1 ml) of the indocyanine green into the ipsilateral upper extremity 10 min before the surgery.
  Near Infra-red images acquisition is performed during surgery
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Subcutaneous injection (1 ml) of the indocyanine green into the ipsilateral upper extremity 10 min before the surgery.
  Near Infra-red images acquisition is performed during surgery

SUMMARY:
The initial standard treatment of breast cancer is surgery. Tumor involvement of lymph nodes is of paramount importance in the subsequent management of this cancer and surgery of invasive breast cancer (BC) involves axillary lymph node dissection (ALND). To preserve arm lymphatic drainage during ALND and avoid the risk of arm lymphedema, mapping the lymphatic drainage by axillary reverse mapping (ARM) has been developed. But oncological safety is uncertain.

The ARM procedure presented here uses indocyanine green (ICG) and fluorescence detection of draining lymphatics. The project aims to train surgeons to the technique and to identify predictive factors for metastatic ARM nodes in invasive BC using tumor and axillary pathological parameters to better select patients who would not require removal of the ARM node in the future

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age
* Preoperative diagnosis of Invasive breast cancer
* Patient deemed for total mastectomy with axillary lymph node dissection (ALND)
* Subject capable of giving informed consent and participating in the process of consent
* Affiliated to the french social security

Exclusion Criteria:

* Mastectomy without ALND
* Previous ipsilateral axillary radiotherapy
* Previous axillary surgery
* Pregnant women as determined by urinary or serum beta human chorionic gonadotropin (hCG) within 72 hours of surgery
* Breastfeeding
* Allergy to indocyanine green
* Patients with a known history of reaction to iodine or iodine-containing compounds.
* No consent
* Impaired capacity to make informed medical decisions
* Patient on guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Rate of identification | up to 30 days
  To determine the Rate of identification of reverse axillary node using Indocyanine green (ICG) and near-infrared (NIR) imaging in invasive breast cancer that undergo total mastectomy and ALND.

CONTACTS AND LOCATIONS:
Overall Officials: Chafika MAZOUNI, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Conversano A, Abbaci M, Karimi M, Mathieu MC, de Leeuw F, Michiels S, Laplace-Builhe C, Mazouni C. Axillary reverse mapping using near-infrared fluorescence imaging in invasive breast cancer (ARMONIC study). Eur J Surg Oncol. 2022 Dec;48(12):2393-2400. doi: 10.1016/j.ejso.2022.07.004. Epub 2022 Jul 8. PMID 35840448
- [Derived] Abbaci M, Conversano A, Karimi M, Mathieu MC, Rouffiac V, De Leeuw F, Michiels S, Laplace-Builhe C, Mazouni C. Near-Infrared Fluorescence Axillary Reverse Mapping (ARM) Procedure in Invasive Breast Cancer: Relationship between Fluorescence Signal in ARM Lymph Nodes and Clinical Outcomes. Cancers (Basel). 2022 May 25;14(11):2614. doi: 10.3390/cancers14112614. PMID 35681595